CLINICAL TRIAL: NCT05403437
Title: Investigation of the Effect of Gestational Diabetes Mellitus on Pelvic Girdle Pain Symptom Severity
Brief Title: Pelvic Girdle Pain Symptom Severity in Pregnant Women With Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 35 09/03/2022
Record Dates: First submitted 2022-04-15; First posted 2022-06-03 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pregnant Women; Gestational Diabetes; Pelvic Girdle Pain
Keywords: pregnant women; pelvic girdle pain; gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational; Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Pregnant women with PGP and newly diagnosed with GDM: Pregnant women with PGP who were newly diagnosed with Gestational Diabetes Mellitus (GDM) according to routine control examinations and whose treatment for diabetes was not started
  Interventions: Other: Evaluation of pain; Diagnostic Test: Evaluation of pelvic girdle pain diagnostic tests; Other: Evaluation of activity limitation
- Group 2: Pregnant women with PGP and diagnosed with GDM: Pregnant women with PGP who were diagnosed with Gestational Diabetes Mellitus (GDM) according to routine control examinations and whose treatment has been already started for diabetes
  Interventions: Other: Evaluation of pain; Diagnostic Test: Evaluation of pelvic girdle pain diagnostic tests; Other: Evaluation of activity limitation
- Group 3: Pregnant women with PGP: Pregnant women with PGP who were not diagnosed with GDM according to routine control examinations
  Interventions: Other: Evaluation of pain; Diagnostic Test: Evaluation of pelvic girdle pain diagnostic tests

INTERVENTIONS:
Other: Evaluation of pain — Painful areas will be marked on the body chart. The presence and severity of pelvic girdle pain will be determined by the Visual Analog Scale (VAS).
Diagnostic Test: Evaluation of pelvic girdle pain diagnostic tests — Pelvic girdle pain diagnostic tests will be applied. The severity of the pain that occurs in positive tests will be evaluated with VAS.
Other: Evaluation of activity limitation — The Pelvic Girdle Questionnaire will be filled.
  Groups: Group 1: Pregnant women with PGP and newly diagnosed with GDM; Group 2: Pregnant women with PGP and diagnosed with GDM

SUMMARY:
Pelvic girdle pain (PGP), which is a common musculoskeletal problem of pregnancy, and gestational diabetes mellitus (GDM), which is diagnosed at the end of the second trimester and at the beginning of the third trimester, occur in a parallel time period. The addition of hyperglycemia to the physiological changes in pregnancy stimulates a new series of cycles and contributes to inflammation, and it is predicted that the presence of GDM may trigger the pain intensity of PGP. Therefore, the aim of this study is to investigate the effect of GDM on PGP symptom severity (pain).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (with PGP) diagnosed with GDM in the 2nd and 3rd trimesters, whose treatment process (diet/insulin) for insulin regulation have been started.
* Pregnant women (with PGP) diagnosed with GDM in the 2nd and 3rd trimesters, whose treatment process (diet/insulin) for insulin regulation have not been started
* Pregnant women (with PGP) who were not diagnosed with GDM in the 2nd and 3rd trimesters

Exclusion Criteria:

* Pre-pregnancy Diabetes Mellitus
* Presence of an orthopedic or neurological problem that may cause musculoskeletal disorders and deviations from normal biomechanical alignment
* Presence of connective tissue disease
* Definition of chronic low back-pelvic region pain (lasting for more than 3 months and pain severity >4 according to VAS) before pregnancy
* History of spine, pelvis, or lower extremity surgery or fracture in the past 6 months
* History of pelvic fracture

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women with PGP and GDM Pregnant women with PGP but without GDM
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Determining of painful areas | Baseline (Current)
  Marking painful areas on the body chart
Evaluation of pain | Baseline (Current)
  Pain will be evaluated with Visual Analog Scale (VAS). The VAS is scaled between 0-10 points (0: no pain, 10: most severe pain).
Application of PGP diagnostic tests | Baseline
  Pelvic Girdle Pain diagnostic tests will be applied. No score defined for test.
Evaluation of PGP severity | Baseline
  The severity of the pain that occurs in positive tests will be evaluated with VAS. The VAS is scaled between 0-10 points (0: no pain, 10: most severe pain).

SECONDARY OUTCOMES:
Pelvic Girdle Questionnaire | Baseline
  Activity limitation will be evaluated Pelvic Girdle Questionnaire
Evaluation of Body Weight | Baseline
  Measuring of the Body Weight
Evaluation of Body Mass Index (BMI) | Baseline
  BMI (kg/m2) will be calculated as person's weight in kilograms divided by the square of height in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aldabe D, Milosavljevic S, Bussey MD. Is pregnancy related pelvic girdle pain associated with altered kinematic, kinetic and motor control of the pelvis? A systematic review. Eur Spine J. 2012 Sep;21(9):1777-87. doi: 10.1007/s00586-012-2401-1. Epub 2012 Jun 21. PMID 22718046
- [Result] Palsson TS, Beales D, Slater H, O'Sullivan P, Graven-Nielsen T. Pregnancy is characterized by widespread deep-tissue hypersensitivity independent of lumbopelvic pain intensity, a facilitated response to manual orthopedic tests, and poorer self-reported health. J Pain. 2015 Mar;16(3):270-82. doi: 10.1016/j.jpain.2014.12.002. Epub 2014 Dec 23. PMID 25540938
- [Result] Plows JF, Stanley JL, Baker PN, Reynolds CM, Vickers MH. The Pathophysiology of Gestational Diabetes Mellitus. Int J Mol Sci. 2018 Oct 26;19(11):3342. doi: 10.3390/ijms19113342. PMID 30373146
- [Result] Eberhard-Gran M, Eskild A. Diabetes mellitus and pelvic girdle syndrome in pregnancy--is there an association? Acta Obstet Gynecol Scand. 2008;87(10):1015-9. doi: 10.1080/00016340802345944. PMID 18763174
- [Result] Wuytack F, O'Donovan M. Outcomes and outcomes measurements used in intervention studies of pelvic girdle pain and lumbopelvic pain: a systematic review. Chiropr Man Therap. 2019 Nov 5;27:62. doi: 10.1186/s12998-019-0279-2. eCollection 2019. PMID 31700607